CLINICAL TRIAL: NCT07400796
Title: Assessing Health System Readiness for Scaling Antenatal MMS in Cambodia: A Mixed-Methods Assessment
Brief Title: Assessing Health System Readiness for Scaling Antenatal MMS in Cambodia
Acronym: TIPS-Cambodia
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Crystal Karakochuk, Associate Professor, Human Nutrition, University of British Columbia
Other Study IDs: TIPSCambodia2026
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Anemia; Pregnancy; Micronutrients; Supplement; Health Systems; Supply Chain Vulnerabilities; Adherence
Keywords: anemia; nutrition; micronutrient; supplement; dietary supplement; Cambodia; policy
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Focus group discussions (FGD) with health centre providers: 15 FGD (5 individuals each)
- Key informant interviews with hospital managers: 17 hospital managers
- Surveys with pregnant individuals who are consuming MMS: 630 pregnant individuals consuming MMS
  Interventions: Dietary Supplement: Multiple micronutrient supplement (MMS) for pregnancy
- Focus group discussion (FGD) with national-level stakeholders in Cambodia: 1 FGD with 5 national-level stakeholders in Cambodia

INTERVENTIONS:
Dietary Supplement: Multiple micronutrient supplement (MMS) for pregnancy — Standard of care MMS during pregnancy (180 tablets total)
  Groups: Surveys with pregnant individuals who are consuming MMS

SUMMARY:
Malnutrition among pregnant women in low- and middle-income countries (LMICs) can cause micronutrient deficiencies that result in adverse maternal and neonatal health outcomes. The World Health Organization has recently recommended antenatal multiple micronutrient supplementation (MMS) that includes iron and folic acid (IFA) to improve maternal and neonatal health outcomes. MMS likely provides additional antenatal benefits over IFA supplementation alone. The Cambodian government, in partnership with Helen Keller International, is piloting MMS implementation in Takeo Province, which will inform nationwide scale-up of MMS.

Study Purpose: The Takeo implementation must be evaluated to understand context-specific implementation of MMS and health system readiness for scale-up. This study assesses system readiness through four domains from the Intervention Scalability Assessment Tool (ISAT): (1) fidelity and adaptation, (2) reach and acceptability, (3) delivery setting and workforce capacity, and (4) implementation infrastructure.

Population: The pilot involves transitioning to MMS from IFA across all 86 health centers, all 6 referral hospitals, and the provincial hospital in Takeo province. This study includes pregnant women receiving antenatal care, antenatal healthcare providers and facilities, and hospital managers in Takeo. The study also includes national governing bodies for MMS delivery.

Methods: This mixed-methods study uses ISAT as a framework for developing data collection methods. Sampling strategies emphasize urban and rural representation across all operational districts in Takeo and diverse stakeholder perspectives at multiple levels of the health system. Data collection includes:

* 12 focus group discussions (FGDs) with health center providers to assess provider adherence to MMS delivery guidelines, perspectives on the transition to MMS, and additional resources needed for MMS delivery
* Workload assessment surveys at FGDs to quantify any burden on providers and resource gaps to deliver MMS
* MMS stockout monitoring at 18 health centers and 7 hospitals to assess supply chain reliability
* 15 key informant interviews with hospital managers to assess perspectives on the integration of MMS into antenatal services and facility readiness for MMS delivery
* Phone surveys with 630 pregnant women to assess acceptability and adherence to MMS at 90- and 180-days after MMS distribution
* One FGD with national-level stakeholders to assess national-level readiness, economic planning, and resource planning for sustainable MMS implementation and scale-up
* Rapid economic evaluation to estimate the cost of nationwide scale-up Potential Impact: This study will generate insights into real-world implementation of MMS in Cambodia. It will identify context-specific adaptations, implementation gaps, and resource planning frameworks needed for nationwide scale-up of MMS. Successful scale-up is anticipated to improve maternal and neonatal health in Cambodia. Findings can also be used to guide other LMICs seeking to transition to and sustainably implement MMS.

ELIGIBILITY:
Inclusion Criteria: For the cohort of pregnant individuals consuming MMS, the inclusion criteria include: 1) current pregnant, 2) at least 18 years of age; 3) have attended at least one ANC visit at a health center or hospital in Takeo during the study period, 4) can provide a functioning phone number for follow-up contact; 5) willingness to participate and provide consent -

Exclusion Criteria: Individuals with diagnosed anemia who require iron and folic acid (IFA) supplementation instead of MMS; (2) individuals unable to communicate via telephone,;(3) individuals who withdraw consent at any point.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 630 individuals will be enrolled in the pregnancy cohort regardless of gestational age to evaluate acceptability and adherence patterns across different pregnancy stages and reflect the real-world setting.
Sampling Method: Non-Probability Sample
Enrollment: 710 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Perspectives on the transition to MMS | 4 months
  12 FGD with health care providers

SECONDARY OUTCOMES:
Additional resources needed for successful MMS delivery | 4 months
  12 FGD with health care providers
Provider adherence to MMS delivery guidelines | 4 months
  12 FGD with health care providers
Adherence of pregnant individuals to MMS supplementation | 6 months
  Adherence, %, of the total 180 tablets prescribed
Perspectives on the integration of MMS into antenatal services and facility readiness for MMS delivery | 4 months
  FGD with hospital managers (key informant interviews)
National-level readiness, economic planning, and resource planning for sustainable MMS implementation and scale-up | 4 months
  FGD with national-level stakeholders
Quantification of any burden on providers and resource gaps to deliver MMS | 4 months
  Workload assessment surveys among the 15 FGD with health center providers

CONTACTS AND LOCATIONS:
Overall Officials: Hou Kroeun, MPH, Study Director — Helen Keller International; Crystal Karakochuk, PHD, Principal Investigator — University of British Columbia; Mai Hoang, MPH, Study Director — Helen Keller International
Locations (1):
- Takeo province, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2026-02-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT07400796/Prot_000.pdf